CLINICAL TRIAL: NCT03452969
Title: Visual Outcomes After Implantation of a Segmental Refractive Multifocal Intraocular Lens Following Cataract Surgery
Brief Title: Visual Outcomes of a Segmental Refractive Multifocal Intraocular Lens
Status: Completed | Type: Observational
Sponsor: University Clinic Frankfurt (Other)
Collaborators: Oculentis GmbH (Unknown)
Responsible Party: Principal Investigator, Myriam Böhm, MD, Professor Dr. med. Thomas Kohnen, University Clinic Frankfurt
Other Study IDs: 153/14
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Visual Acuity
Keywords: visual outcomes; mulitfocal intraocular lens; patient satisfaction; spectacle independence; contrast sensitivity
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Implantation of multifocal intraocular lens — Procedure/Surgery:
  Bilateral implantation of a segmental refractive multifocal intraocular lens (MIOL) following cataract surgery.

SUMMARY:
To evaluate visual outcomes of a segmental refractive multifocal intraocular lens (IOL) after cataract surgery.

DETAILED DESCRIPTION:
Purpose: This prospective, nonrandomized noncomparative case series investigates the visual performance after bilateral implantation of a segmental refractive multifocal intraocular lenses (IOL) after cataract surgery and was performed at the department of Ophthalmology, Goethe University, Frankfurt, Germany.

Methods: Fifty eyes (25 patients) were included. Inclusion criteria were bilateral cataract, age > 45 years, corneal astigmatism ≤ 0.75 D postoperatively, pupil size 3 to 6 mm (mesopic), and center shift < 1 mm (Pentacam). Exclusion criteria were previous ocular surgeries, amblyopia or potential postoperative distance-corrected visual acuity (DCVA) < 0.3 logMAR,

Intervention or Observation: Uncorrected (UCVA) and DCVA in 4 m, 80 cm, 40 cm; contrast sensitivity (CS) under photopic and mesopic conditions; reading skills (Radner Reading Charts); defocus curve, questionnaire on optical quality (OQ) and spectacle independence were assessed after 3 months.

Main Outcome Measures: At 3 months postoperatively, UCVA and DCVA in 4 m, 80 cm, 40 cm (logMAR); defocus curves; CS; reading skills; and OQ questionnaire results.

ELIGIBILITY:
Inclusion Criteria:

* bilateral cataract
* age > 45 years
* corneal astigmatism ≤ 0.75 D postoperatively
* pupil size 3 to 6 mm (mesopic)
* center shift < 1 mm

Exclusion Criteria:

* previous ocular surgeries
* amblyopia
* potential postoperative distance-corrected visual acuity (DCVA) < 0.3 logMAR

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who received bilateral cataract surgery with the implantation of a segmental refractive multifocal intraocular lens
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity at far distance | Measured 3 month after lens surgery
  Monocular and binocular corrected visual acuity at far distance measured in logMAR 3 month after lens surgery

SECONDARY OUTCOMES:
Best corrected visual acuity at intermediate distance | Measured 3 month after lens surgery
  Monocular and binocular corrected visual acuity at intermediate distance measured in logMAR 3 month after lens surgery
Best corrected visual acuity at near distance | Measured 3 month after lens surgery
  Monocular and binocular best corrected visual acuity at near distance measured in logMAR 3 month after lens surgery
Uncorrected visual acuity at far distance | Measured 3 month after lens surgery
  Monocular and binocular uncorrected visual acuity at far distance measured in logMAR 3 month after lens surgery
Uncorrected visual acuity at intermediate distance | Measured 3 month after lens surgery
  Monocular and binocular uncorrected visual acuity at intermediate distance measured in logMAR 3 month after lens surgery
Uncorrected visual acuity at near distance | Measured 3 month after lens surgery
  Monocular and binocular uncorrected visual acuity at near distance measured in logMAR 3 month after lens surgery
Binocular contrast sensitivity (CS) under photopic, mesopic, and mesopic with glare lighting conditions | Measured 3 month after lens surgery
  Binocular contrast sensitivity (CS) was measured with the Functional Acuity Contrast Test (FACT) chart in the Optec 6500 Vision Tester (Stereo Optical Co., Chicago, IL) under binocular photopic (85 cd/m²), mesopic (3 cd/m²), and photopic and mesopic with glare conditions at a spatial frequency of 6 cycles per degree (cpd) (threshold range 0.78-2.26).
Defocus curve testing | Measured 3 month after lens surgery
  Defocus curve (monocular and binocular) was tested from -5.0 D to +2.0 D in 0.5 D steps under photopic lighting conditions (ETDRS).
Radner reading skills | Measured 3 month after lens surgery
  Binocular distance-corrected reading acuity (40 cm) was investigated in LogRAD (Reading Acuity Determination) using reading charts (Radner Reading Charts).
Optical quality questionnaire | Measured 3 month after lens surgery
  Quality of vision questionnaire (visual analogue scale (VAS) 0 (perfect / no symptoms) to 100 (extremely poor / maximum symptom intensity)) asking for evaluation of "glare", "halos", "starbursts", "blurred vision", and "ghosting" under photopic, mesopic and scotopic light conditions, if they wear any spectacles, and to evaluate their total quality of vision.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kohnen, Professor, Principal Investigator — Goethe University Clinic Frankfurt
Locations (1):
- Department of ophthalmology University clinic Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No